CLINICAL TRIAL: NCT05728411
Title: Home Foot-temperature Monitoring Through Smart Mat Technology to Improve Access, Equity, and Outcomes in High-risk Patients With Diabetes
Brief Title: Effectiveness of Remote Foot Temperature Monitoring
Acronym: STOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IIR 21-176
Record Dates: First submitted 2023-02-03; First posted 2023-02-15 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Foot
Keywords: diabetic foot; Dept. of Veterans Affairs; remote sensing technology
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remote temperature monitoring + enhanced usual care (Experimental): Enrollment in remote foot temperature monitoring in addition to enhanced usual care (described below)
  Interventions: Other: Remote foot temperature monitoring system; Other: Enhanced usual care
- Enhanced usual care (Other): Usual care is based on the VA's amputation prevention program (PAVE - Preventing Amputation in Veterans Everywhere - VHA Directive 1410), which provides a model of care for patients at risk for amputation as well as patients who have already undergone an amputation.
  Usual care will be enhanced by providing resources (e.g., information through written newsletters) relevant to a population of Veterans with diabetes, including information on nutrition and cooking, physical activities, and Whole Health opportunities
  Interventions: Other: Enhanced usual care

INTERVENTIONS:
Other: Remote foot temperature monitoring system — Remote temperature monitoring involves a thermometric mat that can detect "hot spots" on the plantar surface of the foot. The mat has embedded cellular connectivity so that data can be transmitted from the patient's home to the company, where the temperature data can be analyzed. The company has a team of health coaches that work with patients and providers to detect signs of damage early in order to prevent ulceration.
  Arms: Remote temperature monitoring + enhanced usual care
Other: Enhanced usual care — Usual care is based on the VA's amputation prevention program (PAVE - Preventing Amputation in Veterans Everywhere - VHA Directive 1410), which provides a model of care for patients at risk for amputation as well as patients who have already undergone an amputation.
  Usual care will be enhanced by providing resources (e.g., information through written newsletters) relevant to a population of Veterans with diabetes, including information on nutrition and cooking, physical activities, and whole health opportunities

SUMMARY:
Diabetic foot ulcers are common, debilitating, and costly complications of diabetes, disproportionately impacting Black and rural Veterans. Forty percent of individuals have an ulcer recurrence within a year of ulcer healing and 65% within 5 years. Monitoring plantar foot temperatures is one of the few interventions that reduces the risk of ulcer recurrence. Despite the evidence, adoption has been poor because the original procedures, including the use of handheld thermometers, were burdensome and time-consuming. Podimetrics, a private company, has developed a temperature monitoring system involving a "smart" mat that can wirelessly transmit data and a remote monitoring team that works with VA providers to assist with triage and monitoring. This care model has incredible promise, but has been untested in VA. The investigators propose to conduct a randomized trial to evaluate effectiveness of remote temperature monitoring as well as costs. Additionally, the investigators will evaluate the implementation process, including barriers and facilitators to use among key stakeholders.

DETAILED DESCRIPTION:
Objective(s) and Hypotheses: Diabetic foot ulcers (DFU) are common, debilitating, and costly complications of diabetes, disproportionately impacting Black and rural Veterans. Forty percent of individuals have an ulcer recurrence within a year of ulcer healing and 65% within 5 years. Remote temperature monitoring (RTM) of feet is one of the few interventions that reduces the risk of ulcer recurrence. Despite the evidence, adoption has been poor because the original procedures, including the use of handheld thermometers, were burdensome and time-consuming. Podimetrics, a private company, has developed a temperature monitoring system involving a "smart" mat that measure foot temperatures and a remote monitoring team that works with VA providers to assist with triage and monitoring. This care model has incredible promise, but has been untested in VA.

The specific aims of this study are to: 1) Evaluate the effectiveness of RTM vs. usual care in terms of primary (ulceration) and secondary outcomes (severity of ulceration, amputation, hospitalization, emergency room visits, quality of life, satisfaction with care, and self-efficacy for managing diabetes) at 6, 12, 18, and 24 months; 2) Collect data on costs of RTM and compare with usual care costs, if effectiveness is demonstrated; and 3) Evaluate the implementation process, including barriers and facilitators to use among key stakeholders

Research Design: For Aim 1, the investigators will conduct a multi-site randomized controlled study. Aim 2 involves a budget impact analysis to evaluate costs of RTM. Aim 3 involves qualitative interviews to understand barriers and facilitators to implementation of RTM.

Methodology: For Aim 1, the investigators will aim to enroll at least 406 patients who have had a history of DFU or amputation (including active ulcers). Patients will be randomized 1:1 to RTM or usual care (no RTM), with randomization stratified on site and active ulcer vs. not. For Aim 2, the investigators will collect data and observe providers to quantify provider time for selecting patients for RTM, ordering mats, and responding to alerts of "hot spots". The investigators will use medical records to assess patient utilization (ulcer/amputation-related outpatient, inpatient, and emergency room visits) and associated costs of care for patients in the RTM and comparison groups. For Aim 3, the investigators will conduct semi-structured phone interviews with 30-50 Veterans and 12-30 providers and use the Consolidated Framework for Implementation Research to guide data collection and analysis.

Relevance to VA Mission: Findings from this study will be used to inform effective, efficient, and equitable scaling of RTM in VA.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Diabetes diagnosis
* History of foot ulcer (including active ulcer) OR history of lower extremity amputation (including unhealed amputation)
* Able to understand/read English

Exclusion Criteria:

* Dementia
* Unable to ambulate
* Bilateral lower extremity amputation
* Ankle brachial index <0.6 or toe brachial index <0.5
* Currently using in-home temperature monitoring
* Prisoner

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of foot ulceration | 24 months
  The primary outcome is the presence of new ulceration through 24 months

SECONDARY OUTCOMES:
Rate of lower limb amputation | 24 months
  Any level of lower extremity amputation
Mean or median quality of life scores | 6,12, 18 and 24 months
  Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health v1.2. The global scale produces two scores: Global Mental Health and Global Physical Health. Raw scores are converted to T-score values (higher values indicate better health). Minimum and maximum T scores for Global Mental Health are 21.2 and 67.6, respectively. Minimum and maximum T scores for Global Physical Health are 16.2 and 67.7, respectively.
Mean or median satisfaction with care scores | 6,12, 18 and 24 months
  Short assessment of patient satisfaction (SAPS) by Hawthorne G et al (2006) which includes 7 items. Each item is scored on a 0 to 4 scale. The score range is from 0 (extremely dissatisfied) to 28 (extremely satisfied).
Mean or median self-efficacy for diabetes | 6, 12, 18, and 24 months
  8-item Self-efficacy for diabetes measure that has a range of 1 to 10. Higher scores indicate higher self-efficacy.

OTHER OUTCOMES:
Utilization (outpatient visits, emergency room visits, hospitalizations) - any vs. none and number | 6, 12, 18, and 24 months
  Based on electronic medical record data

CONTACTS AND LOCATIONS:
Overall Officials: Alyson J. Littman, PhD MPH, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (4):
- United States (4):
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Richmond VA Medical Center, Richmond, VA, Richmond, Virginia
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington
  - Spokane VA Medical Center, Spokane, WA, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No
Subject to IRB approval, de-identified data will be released to a local VAPSHCS and/or national VA research data repository for release to non-VA protocols. The VA research data repository administrator will be responsible for reviewing and responding to requests to release data to non-VA requesters. A data use agreement compliant with VHA Handbooks 1200.12 and 1605.1 will be required between VHA and the requester. Review and approval by VA privacy officer is required prior to disclosure.